CLINICAL TRIAL: NCT01223560
Title: Collection of Information-Rich Type 1 Diabetes Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: The Danish Council for Strategic Research (Other); Technical University of Denmark (Other); Novo Nordisk A/S (Industry)
Responsible Party: Signe Schmidt, MD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: DiaCon Study 01
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Type 1 Diabetes
Keywords: Artificial pancreas; Model predictive control; Virtual patient
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Exercise; Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Insulin Aspart — Insulin bolus with and without carbohydrate intake.
Other: Exercise — Exercise on tread mill
Dietary Supplement: Carbohydrate — Carbohydrate intake

SUMMARY:
The aim of this clinical study was to obtain type 1 diabetes data to identify models for glucose prediction and control and to construct a physiological pharmaco-kinetic/pharmaco-dynamic computer model of a type 1 diabetic person.

ELIGIBILITY:
Inclusion Criteria:

* diabetes duration > 5 years
* HbA1c < or = 7.2%
* CSII treated for > 3 months
* Capable of being moderately, physically active for 20 minutes

Exclusion Criteria:

* symptoms of diabetic late complications except simplex retinopathy
* pregnancy or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark